CLINICAL TRIAL: NCT04066426
Title: Analgesic Efficacy of Naproxen-codeine, Naproxen+Dexamethasone, and Naproxen on Myofascial Pain: A Randomized Double-blind Controlled Trial
Brief Title: Efficacy of Naproxen-codeine, Naproxen+Dexamethasone, and Naproxen on Myofascial Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, levent Cigerim, Head of Oral and Maxillofacial Surgery Department, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16.02.2018/12
Record Dates: First submitted 2019-08-17; First posted 2019-08-26 (Actual); Results first posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-01

CONDITIONS: Temporomandibular Disorder
Keywords: naproxen sodium; codeine phosphate; dexamethasone; pain; temporomandibular joint
MeSH Terms: conditions — Temporomandibular Joint Disorders; Pain | interventions — Naproxen; Acetaminophen; Codeine; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- naproxen sodium+codeine phosphate (Experimental): Naproxen sodium is a propionic acid derivative with analgesic, antipyretic, and antiinflammatory properties. Its mechanism of action relies on the inhibition of prostaglandin synthesis, and significant pain relief and plasma levels can be obtained within 20 minutes following intake. The elimination half-life of naproxen sodium is reportedly around 14 hours, and naproxen sodium is used in doses ranging from 275 to 550 mg in surgical procedures. Codeine phosphate is an opioid analgesic which has similar applications to those of morphine. However, it is significantly less potent as an analgesic and has only mild sedative effects. The drug's principal site of action is at the µ-opioid receptors (MOR) which are distributed in the central nervous system. Peak effect is reached within 2 hours and analgesic action continues for approximately 4 hours. Naproxen sodium (550 mg)+codeine phosphate (30 mg) was used twice daily in this study.
  Interventions: Drug: naproxen sodium+codeine phosphate, naproxen sodium+dexamethasone, naproxen sodium, paracetamol
- naproxen sodium+dexamethasone (Experimental): Naproxen sodium is a propionic acid derivative with analgesic, antipyretic, and antiinflammatory properties. Its mechanism of action relies on the inhibition of prostaglandin synthesis, and significant pain relief and plasma levels can be obtained within 20 minutes following intake. The elimination half-life of naproxen sodium is reportedly around 14 hours, and naproxen sodium is used in doses ranging from 275 to 550 mg in surgical procedures. Naproxen sodium (550 mg) was used twice daily + dexamethasone (8 mg) was used once daily in this study.
  Interventions: Drug: naproxen sodium+codeine phosphate, naproxen sodium+dexamethasone, naproxen sodium, paracetamol
- naproxen sodium (Experimental): Naproxen sodium is a propionic acid derivative with analgesic, antipyretic, and antiinflammatory properties. Its mechanism of action relies on the inhibition of prostaglandin synthesis, and significant pain relief and plasma levels can be obtained within 20 minutes following intake. The elimination half-life of naproxen sodium is reportedly around 14 hours, and naproxen sodium is used in doses ranging from 275 to 550 mg in surgical procedures. Naproxen sodium (550 mg) was used twice daily in this study.
  Interventions: Drug: naproxen sodium+codeine phosphate, naproxen sodium+dexamethasone, naproxen sodium, paracetamol
- paracetamol (Active Comparator): Paracetamol is a mild analgesic and antipyretic, and is recommended for the treatment of most painful and febrile conditions, for example, headache including migraine, toothache, neuralgia, colds and influenza, sore throat, backache, rheumatic pain and dysmenorrhoea.
  Interventions: Drug: naproxen sodium+codeine phosphate, naproxen sodium+dexamethasone, naproxen sodium, paracetamol

INTERVENTIONS:
Drug: naproxen sodium+codeine phosphate, naproxen sodium+dexamethasone, naproxen sodium, paracetamol — NSAID, steroid, opioid, paracetamol and combinations of this drugs can be used in temporomandibular disorders.
  Other Names: Anaprox Double Strength (DS) + Codeine, Anaprox DS + Decadron, Anaprox DS, Parmol

SUMMARY:
Temporomandibular disorders (TMDs) are one of the most common muco-skeletal disorders, seen in the dental clinics. Many factors work together to initiate or aggravate the condition, so it is a multifactorial disorder. The etiology of TMDs may be a result of parafunctional habits such as clenching and bruxism, acute trauma to the jaw, trauma from hyperextension e.g. after a long dental treatment, joint laxity, psychological distress, occlusal disharmony like presence of high crown or free-end saddle leading to joint instability or systemic diseases such as Rheumatoid arthritis or Osteoarthritis. The aim of this study was to evaluate the effects of naproxen sodium+codeine phosphate, naproxen sodium+dexamethasone, and naproxen sodium on pain in patients complaining from temporomandibular pain.

ELIGIBILITY:
Inclusion Criteria:

* Without a systemic disease,
* Not used any medication in the last week
* Have a habit of clenching and / or grinding teeth, individuals with normal preoperative results, suffering with pain and / or limitation of the mouth opening in the temporomandibular region

Exclusion Criteria:

Individuals who smoke

* Have a parafunctional habits (except for squeezing and grinding teeth)
* Pregnant and breastfeeding individuals
* Allergies to study medicines
* Do not use their medications / use different drugs and non-follow-up

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Volkan KAPLAN, PhD, Study Chair — Cairo University
Locations (1):
- Van Yuzuncu Yil University, Faculty of Dentistry, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naproxen Sodium+Codeine Phosphate | Naproxen Sodium+Dexamethasone | Naproxen Sodium | Paracetamol
Started | 50 | 50 | 50 | 50
Completed | 40 | 40 | 42 | 47
Not Completed | 10 | 10 | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naproxen Sodium+Codeine Phosphate | Naproxen Sodium+Dexamethasone | Naproxen Sodium | Paracetamol | Total
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Thirty-one patients were excluded from the study due to 26 patients having been lost to follow-up, 2 patients used different medication, and 3 patients did not comply with the intended drug dosage.
  years
    number analyzed (Participants) | 40 | 40 | 42 | 47 | 169
    (all) | 26.18 (10.06) | 27.15 (10.86) | 29.38 (11.72) | 25.60 (9.57) | 27.04 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Thirty-one patients were excluded from the study due to 26 patients having been lost to follow-up, 2 patients used different medication, and 3 patients did not comply with the intended drug dosage.
  Participants
    number analyzed (Participants) | 40 | 40 | 42 | 47 | 169
    Female | 33 | 28 | 36 | 35 | 132
    Male | 7 | 12 | 6 | 12 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pain Evaluation
Description: Evaluation of changes in Visual Analog Scale measurements by groups (0 = no pain; 10 = unbearable pain)
Time Frame: Pre-treatment (baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naproxen Sodium+Codeine Phosphate | Naproxen Sodium+Dexamethasone | Naproxen Sodium | Paracetamol
Number analyzed (Participants) | 40 | 40 | 42 | 47
score on a scale | 6.38 (1.86) | 6.93 (1.76) | 5.76 (2.74) | 5.49 (2.73)

2. Primary Outcome: Pain Evaluation
Description: Evaluation of changes in Visual Analog Scale measurements by groups (0 = no pain; 10 = unbearable pain).
Time Frame: At the first week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naproxen Sodium+Codeine Phosphate | Naproxen Sodium+Dexamethasone | Naproxen Sodium | Paracetamol
Number analyzed (Participants) | 40 | 40 | 42 | 47
score on a scale | 4.68 (1.82) | 5.93 (2.22) | 4.95 (2.85) | 4.60 (2.89)

3. Primary Outcome: Pain Evaluation
Description: Evaluation of changes in Visual Analog Scale measurements by groups (0 = no pain; 10 = unbearable pain).
Time Frame: At the second week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naproxen Sodium+Codeine Phosphate | Naproxen Sodium+Dexamethasone | Naproxen Sodium | Paracetamol
Number analyzed (Participants) | 40 | 40 | 42 | 47
score on a scale | 3.58 (1.69) | 5.28 (2.36) | 4.33 (2.78) | 4.34 (3.03)

4. Primary Outcome: Pain Evaluation
Description: Evaluation of changes in Visual Analog Scale measurements by groups (0 = no pain; 10 = unbearable pain).
Time Frame: At the first month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naproxen Sodium+Codeine Phosphate | Naproxen Sodium+Dexamethasone | Naproxen Sodium | Paracetamol
Number analyzed (Participants) | 40 | 40 | 42 | 47
score on a scale | 2.93 (1.65) | 5.28 (2.50) | 3.69 (2.71) | 4.38 (2.96)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Naproxen Sodium+Codeine Phosphate | Naproxen Sodium+Dexamethasone | Naproxen Sodium | Paracetamol
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/42 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/42 | 0/47
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/42 | 0/47

LIMITATIONS AND CAVEATS:
The diversity of the individuals in the groups was the limitation of this study. Different individual characteristics may change the efficacy of drugs in groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT04066426/Prot_SAP_000.pdf